CLINICAL TRIAL: NCT02110355
Title: A Phase 1b/2a Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of AMG 232 Combined With Trametinib and Dabrafenib or Trametinib in Adult Subjects With Metastatic Cutaneous Melanoma
Brief Title: A Phase 1b/2a Study Evaluating AMG 232 in Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120238
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Oncology; Oncology Patients; Tumors; Melanoma
Keywords: Metastatic melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; trametinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AMG 232 with Trametinib and Dabrabenib (Experimental): Arm 1 of Part 1 and 2 and Part 3
  Interventions: Drug: AMG 232; Drug: Trametinib; Drug: Dabrafenib
- AMG 232 with Trametinib (Experimental): Arm 2 of Part 1 and 2
  Interventions: Drug: AMG 232; Drug: Trametinib
- Trametinib and Dabrafenib (Active Comparator): Part 3
  Interventions: Drug: Trametinib; Drug: Dabrafenib

INTERVENTIONS:
Drug: AMG 232 — Given as an oral tablet in escalating doses
  Arms: AMG 232 with Trametinib; AMG 232 with Trametinib and Dabrabenib
Drug: Trametinib — Trametinib is an anti-cancer agent
Drug: Dabrafenib — Dabrafenib is an anti-cancer agent
  Arms: AMG 232 with Trametinib and Dabrabenib; Trametinib and Dabrafenib

SUMMARY:
Phase 1b/2a, open-label, sequential dose escalation and expansion study of AMG 232 in combination with trametinib and dabrafenib in subjects with metastatic melanoma followed by a direct comparison of AMG 232 combined with trametinib and dabrafenib versus trametinib combined with dabrafenib alone.

DETAILED DESCRIPTION:
The study will be conducted in 3 parts: Part 1 - Dose Escalation, Part 2 - Dose Expansion and Part 3, a randomized Phase 2a.

In both part 1 and 2, subjects will be enrolled open-label into 1 of 2 arms. For both Arm 1 and Arm 2, the part 1 dose escalation is aimed at determining an AMG 232 maximum tolerated dose (MTD) with a fixed dose of the combination drug(s) and evaluating safety, tolerability, pharmacokinetics and pharmacodynamics of each combination. Part 2 dose expansion will enroll subjects to receive therapy with a dose and schedule of AMG 232 selected from the corresponding part 1 dose escalation. In part 2 subjects will be enrolled to confirm safety and tolerability and to assess clinical activity prior to proceeding to Part 3, Phase 2a. In Phase 2a, Subjects will be randomized open-label in a 1:1 ratio to receive AMG 232 in combination with trametinib plus dabrafenib versus trametinib plus dabrafenib alone.

Only Part 1 of the study was enrolled and the study did not proceed into Phase 2.

ELIGIBILITY:
Inclusion Criteria: Subjects must have histologically or cytologically confirmed metastatic cutaneous or mucosal melanoma, Able to swallow and retain orally administered medication, Adequate hematological, renal, hepatic, and coagulation laboratory assessments Exclusion Criteria: Clinically significant bleeding within 4 weeks of screening, Current use of warfarin, factor Xa inhibitors, and direct thrombin inhibitors, Infection requiring anti-infective treatments within 1 week of study enrollment, Anti-tumor therapy, Major surgery within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events, Results of safety laboratory tests, vital sign measurements, ECG measurements, PK parameters; Progression-free Survival Rate | 36 months
  Incidence and grade of treatment-emergent adverse events, including dose-limiting toxicities; AMG 232, trametinib, dabrafenib, and metabolite PK parameters; progression-free Survival

SECONDARY OUTCOMES:
Time to and duration of overall response and duration of stable disease measured by CT or MRI and assessed per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, Progression-free and Overall Survival | 36 months
  Objective Tumor Response

CONTACTS AND LOCATIONS:
Overall Officials: John Mei, Study Director — Kartos Therapeutics
Locations (7):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Nashville, Tennessee
- Australia (2):
  - Research Site, North Sydney, New South Wales
  - Research Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No